CLINICAL TRIAL: NCT05502146
Title: Comparison of Two Different Norepinephrine Bolus Doses for Management of Spinal Anesthesia-Induced Hypotension in Cesarean Section: A Randomized Controlled Study
Brief Title: Comparison of Two Different Norepinephrine Bolus Doses for Management of Spinal Anesthesia-Induced Maternal Hypotension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Assistant Prof Levent Özdemir, M.D., Assistant Professor, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022/05
Record Dates: First submitted 2022-08-10; First posted 2022-08-16 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Spinal Anesthetic Toxicity; Hypotension Drug-Induced; Cesarean Section Complications
MeSH Terms: conditions — Hypotension | interventions — Norepinephrine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bolus 6 micrograms Noradrenaline group (Experimental): Mothers in this group will receive a bolus of Norepinephrine 6 mcg for management of hypotensive episode after spinal anesthesia using Bupivacaine hydrochloride.
  Interventions: Drug: Noradrenaline Bitartrate; Drug: Bupivacaine Hydrochloride
- Bolus 8 micrograms Noradrenaline group (Active Comparator): Mothers in this group will receive a bolus of Norepinephrine 8 mcg for management of hypotensive episode after spinal anesthesia using Bupivacaine hydrochloride.
  Interventions: Drug: Noradrenaline Bitartrate; Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Noradrenaline Bitartrate — An intravenous bolus of norepinephrine 6 mcg will be administered for management of maternal hypotension.
  Other Names: Stenor
  Arms: Bolus 6 micrograms Noradrenaline group
Drug: Bupivacaine Hydrochloride — Subarachnoid block will be performed using Bupivacaine hydrochloride (2.5 mL)
  Other Names: Marcaine Spinal Heavy
  Arms: Bolus 6 micrograms Noradrenaline group
Drug: Noradrenaline Bitartrate — An intravenous bolus of norepinephrine 8 mcg will be administered for management of maternal hypotension.
  Other Names: Stenor
  Arms: Bolus 8 micrograms Noradrenaline group
Drug: Bupivacaine Hydrochloride — Subarachnoid block will be performed using Bupivacaine hydrochloride (2.5 mL)
  Other Names: Marcaine Spinal Heavy
  Arms: Bolus 8 micrograms Noradrenaline group

SUMMARY:
In this study the investigators will compare two doses of norepinephrine bolus (6 mcg and 8 mcg) in management of maternal hypotensive episode after spinal block during cesarean delivery.

DETAILED DESCRIPTION:
Maternal hypotension after spinal anesthesia is a common and serious complication during cesarean delivery. Despite all preventive measures, the incidence of hypotension is still around 20%. In these cases, maternal hypotension treatment is usually required using vasopressor boluses. One of the vasopressors commonly used during cesarean delivery is norepinephrine, especially recently.

Although phenylephrine has long been the first choice for the prevention and treatment of maternal hypotension, its use may cause bradycardia and decreased maternal cardiac output.

Norepinephrine is an alpha adrenergic agonist with weak beta adrenergic agonistic activity; therefore, it does not cause significant cardiac depression like phenylephrine. Norepinephrine has been introduced for use during cesarean delivery with promising results. Several previous studies have investigated the efficacy of norepinephrine infusion in preventing maternal hypotension. A dose-response study investigated the best dose of Norepinephrine for the prevention of hypotension. In the dose-response study mentioned above, a dose of 6 mcg was reported as the best dose for prophylaxis against hypotension.

There are very limited studies investigating the best bolus dose of norepinephrine for the treatment of maternal hypotensive episode, and the optimal dose recommendation is uncertain. In this study, researchers will investigate the efficacy and adverse effects of two bolus doses of norepinephrine (6 mcg and 8 mcg) in the management of a maternal hypotensive episode after subarachnoid block during cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Woman,
* ASA I-II,
* 18-49 age range,
* Actual body weight >50 kg,<90 kg
* Actual height >150cm, <180cm
* Patients undergoing surgery under elective conditions and emergency cases for non-bleeding reasons
* Fasting period is appropriate,
* Term pregnancy (38-42 weeks),
* Patients without cardiovascular disease
* Spinal block that does not reach the high level (<T4),
* Patients without diagnosis of stage 2 or higher hypertension hypertension (Stage 2 hypertension is defined as a systolic blood pressure of more than 160 mmHg and a diastolic blood pressure of more than 90 mmHg.),
* Patients without vasoactive drug use,
* Preop Systolic Blood Pressure >90 mmHg,
* Bleeding less than 750 ml,
* Patients who signed the informed consent form to be included in the study

Exclusion Criteria:

* ASA III-IV,
* Pregnant women outside the age range of 18-49,
* Actual body weight >90kg, <50kg
* Actual height >180cm, <150cm
* Patients with inappropriate fasting time
* Preterm pregnancy (<38 weeks) or postterm pregnancy (>42 weeks)
* Bleeding amount more than 750 ml
* Emergency surgery with bleeding (previa, placental abruption, etc.)- Pregnant with cardiovascular system disease,
* High block level (>T4)
* Having a diagnosis of stage 2 or higher hypertension hypertension (Stage 2 hypertension is defined as a systolic blood pressure of more than 160 mmHg and a diastolic blood pressure of more than 90 mmHg.),
* Use of vasoactive drugs,
* Preop Systolic Blood Pressure <90 mmHg
* Patients who did not sign the informed consent form to be included in the study

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female patients with cesarean delivery
Enrollment: 200 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Rate of successful management of maternal hypotension | After spinal anesthesia until the end of surgery
  Number of patients with successful management of a maternal hypotensive episode (defined as systolic blood pressure greater than 80% of baseline measurement and systolic blood pressure greater than 90 mmHg) Successful management is considered to be successful management if blood pressure does not fall below 90 mmHg and 80% of baseline measurement within 6 minutes after norepinephrine administration after hypotension develops.
Number of Noradrenaline doses administered and total dose amount | After spinal anesthesia until the end of surgery
  Evaluation of the number of bolus noradrenaline doses and the total dose required for the treatment of maternal hypotension after spinal block.

SECONDARY OUTCOMES:
Incidence of reactive hypertension | After spinal anesthesia until the end of surgery
  Number of patients with reactive hypertension (defined as systolic blood pressure ≥120% from the baseline reading after administration of norepinephrine bolus).
Incidence of bradycardia | After spinal anesthesia until the end of surgery
  Patients with a heart rate less than 40 bpm
Evaluation of "Appearance, Pulse, Grimace, Activity, and Respiration" (APGAR) score | The first 5 minutes after birth
  The minimum score that can be obtained from this scale is 0 and the maximum is 10 points.
  Scoring will be calculated at 1 and 5 minutes immediately after birth. A score of 9 to 10 is consistent with a better clinical outcome, while a score of 8 or less will be considered a poor clinical outcome.
Umbilical cord blood gas analyses of fetus | The first 5 minutes after birth
  Potential of hydrogen (pH): Normal range is between 7.35-7.45
Umbilical cord blood gas analyses of fetus | The first 5 minutes after birth
  Partial arterial oxygen pressure (PaO2, mmHg): Normal range is between 50-100 mmHg
Umbilical cord blood gas analyses of fetus | The first 5 minutes after birth
  Partial carbon dioxide pressure (PaCO2, mmHg): Normal range is between 35-45 mmHg
Umbilical cord blood gas analyses of fetus | The first 5 minutes after birth
  Bicarbonate (HCO3, mEq/liter): Normal range is between 22-26 mEq/liter
Umbilical cord blood gas analyses of fetus | The first 5 minutes after birth
  Base deficit (BE, mEq/liter): Normal range is between +2 to -2 mEq/liter
The frequency of side effects after norepinephrine | During surgery after spinal block
  the number of patients with side effects (Nausea, vomiting, headache, tinnitus, arrhythmia, chest pain, etc.)
The frequency of side effects after subarachnoid block | During surgery after spinal block
  Side effects seen after spinal block and in patients who have not yet received noradrenaline
Effect of noradrenaline on heart rate variability | Measurements just before and 1 minute after noradrenaline administration
  Comparison of the rates of change in heart rate in measurements before and after two different bolus doses of noradrenaline.

CONTACTS AND LOCATIONS:
Overall Officials: Levent Özdemir, Assist Prof, Principal Investigator — Mersin University
Locations (1):
- Mersin University, Mersin, Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Onwochei DN, Ngan Kee WD, Fung L, Downey K, Ye XY, Carvalho JCA. Norepinephrine Intermittent Intravenous Boluses to Prevent Hypotension During Spinal Anesthesia for Cesarean Delivery: A Sequential Allocation Dose-Finding Study. Anesth Analg. 2017 Jul;125(1):212-218. doi: 10.1213/ANE.0000000000001846. PMID 28248702
- [Background] Chen D, Qi X, Huang X, Xu Y, Qiu F, Yan Y, Li Y. Efficacy and Safety of Different Norepinephrine Regimens for Prevention of Spinal Hypotension in Cesarean Section: A Randomized Trial. Biomed Res Int. 2018 May 23;2018:2708175. doi: 10.1155/2018/2708175. eCollection 2018. PMID 29951531
- [Background] Carvalho B, Dyer RA. Norepinephrine for Spinal Hypotension during Cesarean Delivery: Another Paradigm Shift? Anesthesiology. 2015 Apr;122(4):728-30. doi: 10.1097/ALN.0000000000000602. No abstract available. PMID 25654435
- [Result] Hassabelnaby YS, Hasanin AM, Adly N, Mostafa MMA, Refaat S, Fouad E, Elsonbaty M, Hussein HA, Mahmoud M, Abdelwahab YM, Elsakka A, Amin SM. Comparison of two Norepinephrine rescue bolus for Management of Post-spinal Hypotension during Cesarean Delivery: a randomized controlled trial. BMC Anesthesiol. 2020 Apr 17;20(1):84. doi: 10.1186/s12871-020-01004-y. PMID 32303180